CLINICAL TRIAL: NCT07314658
Title: The Effects of Time-restricted Eating (TRE) With and Without Additional Protein on Body Composition, Muscle Function and Markers of Metabolic Health in Older Adults
Brief Title: Time-restricted Eating (TRE) and Protein in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 361019
Record Dates: First submitted 2025-11-26; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Generally Healthy Adults Over 60 Years Old
MeSH Terms: interventions — Trehalase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TRE (Experimental): Participants undertaking the TRE intervention
  Interventions: Other: TRE
- ProtAM TRE (Experimental): Participants undertaking the ProtAM TRE intervention
  Interventions: Other: ProtAM TRE
- ProtPM TRE (Experimental): Participants undertaking the ProtPM TRE intervention
  Interventions: Other: ProtPM TRE
- Control (No Intervention)

INTERVENTIONS:
Other: TRE — * Participants will be asked to follow a 16:8 TRE protocol, consuming all their daily within 8 hours, between 12 and 8pm, and fast for 16 hours overnight.
  * Outside of the eating window, participants will be allowed to consume energy-free drinks only, i.e. water, black tea/coffee, 0-calorie soft drinks.
  Arms: TRE
Other: ProtAM TRE — * Participants will be asked to follow a 16:8 TRE protocol, consuming all their daily within 8 hours, between 12 and 8pm, and fast for 16 hours overnight.
  * Outside of the eating window, participants will be allowed to consume energy-free drinks only, i.e. water, black tea/coffee, 0-calorie soft drinks.
  * In addition, they will be asked to consume a protein drink containing 30g protein in the morning, 2 hours before the 8-hour eating window opens at 12pm (i.e. at 10am).
  Other Names: TRE + morning protein 'snack'
  Arms: ProtAM TRE
Other: ProtPM TRE — * Participants will be asked to follow a 16:8 TRE protocol, consuming all their daily within 8 hours, between 12 and 8pm, and fast for 16 hours overnight.
  * Outside of the eating window, participants will be allowed to consume energy-free drinks only, i.e. water, black tea/coffee, 0-calorie soft drinks.
  * In addition, they will be asked to consume a protein drink containing 30g protein in the afternoon, either 2 hours after their first meal or 2 hours before their last meal of the day.
  Other Names: TRE + afternoon protein 'snack'
  Arms: ProtPM TRE

SUMMARY:
The aim this study is to investigate the effects of time-restricted eating (TRE) on body composition, muscle function and markers of metabolic health of adults over 60 years old. This study will compare different variations of TRE - with and without an additional protein.

This study involves attending two study days at the University of Surrey for baseline and end-of-intervention measurement of body composition using a gold-standard dual energy x-ray absorptiometry (DEXA) scan; muscle function using hand grip strength and 30-second sit-to-stand tests; weight. A blood sample will be taken at each study visit to measure markers of lipid and glucose control, and insulin sensitivity.

Participants will be randomly allocated to one of four study groups:

* control group: maintain habitual dietary patterns
* TRE group: fast for 16 hours overnight, eat between 12-8pm
* TRE + Protein (AM): fast for 16 hours overnight, eat between 12-8pm; take a 30g plant-based protein supplement in the morning
* TRE + Protein (PM): fast for 16 hours overnight, eat between 12-8pm; take a 30g plant-based protein supplement in the afternoon Participants will be asked to follow the intervention according to their allocated group for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female
* Age range: 60 years or older
* Fasting for 12 or less hours on a daily basis
* BMI range: 23-30 kg/m2
* Weight stability: no more than 3kg weight gain or loss in the past 3 months
* Regular eating pattern, i.e. 3 meals a day
* Able to prepare the protein supplement

Exclusion Criteria:

* Any of the following present (in line with exclusion criteria used in previous TRE research in older adults):

  * known renal impairment
  * heart attack or stroke in the past three months
  * continuous use of supplemental oxygen to manage a chronic pulmonary condition or heart failure
  * rheumatoid arthritis
  * Parkinson's disease
  * active treatment for cancer in the past year
  * insulin dependent diabetes mellitus
* taking medications that preclude fasting for 16 h
* actively trying or planning to lose weight
* history of an eating disorder
* outside of stated age or BMI range
* fasting for longer than 12 hours on a daily basis
* unable to prepare the protein supplement
* extreme morning/evening chronotype
* sleep disorders
* regular meal skipping
* history of difficulty having a blood sample taken
* Recent exposure to high-dose radiation
* Vigorous exercise on more than 3 occasions a week

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body composition at 2 months using whole-body dual-energy x-ray absorptiometry (DEXA) | For 8 weeks of the assigned study intervention
  Measured using whole-body dual-energy x-ray absorptiometry (DEXA) In addition to the above, body composition will also be assessed using Tanita Bioelectrical impedance analysis (BIA). Fat free and fat mass will be reported in kg.
Change from baseline in muscle function at 2 months | At the start and end of 8 weeks of the assigned study intervention
  Measured using grip strength
Change from baseline in muscle function at 2 months | At the start and end of 8 weeks of the assigned study intervention
  Measured using 30-second sit-to-stand test.

SECONDARY OUTCOMES:
Change in fasting glucose control indicators | At the start and end of 8 weeks of the assigned study intervention
  HbA1c
Change from baseline in insulin sensitivity at 2 months | At the start and end of 8 weeks of the assigned study intervention
  HOMA-IR
Change from baseline in lipid metabolism at 2 months | At the start and end of 8 weeks of the assigned study intervention
  fasting total, LDL- and HDL cholesterol and triglyerides
Change from baseline in diet composition at 2 months | At the start, mid-point (week 4) and end of 8 weeks of the assigned study intervention
  Macro- and micronutrient analysis using the nutrition analysis platform Nutritics of 3-day food diaries administered at the start, mid-point and end of the assigned study intervention.
Feasibility of the assigned TRE intervention | at the end of the 8 week intervention
  semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not required or applicable for this study protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT07314658/Prot_SAP_000.pdf